CLINICAL TRIAL: NCT00213083
Title: Phase 3 Study of the Efficacy and Safety of the Microbicide Carraguard® in Preventing HIV Seroconversion in Women
Brief Title: Efficacy Study of the Vaginal Gel Carraguard to Prevent HIV Transmission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Population Council #322
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections; AIDS; Sexually Transmitted Diseases; HIV Seroconversion
Keywords: Microbicide; HIV; AIDS; STIs; STDs; Efficacy; HSV; Women; South Africa; seroconversion; condom; safe-sex; vaginal intercourse; prevention; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; HIV Seropositivity; Safe Sex; Coitus

INTERVENTIONS:
Drug: Carraguard (PC-515)

SUMMARY:
The purposes of this study are to determine whether Carraguard® Gel can prevent the transmission of HIV when used during vaginal intercourse, and to confirm that the gel is safe for vaginal use.

DETAILED DESCRIPTION:
This study is designed to show if Carraguard® can protect women against HIV if it is used before sex, and is safe for long-term use.

ELIGIBILITY:
Inclusion Criteria:

* HIV negative and agree to be tested for HIV and told their results at all visits during the study
* Aged 16 - 40 years of age
* Have had at least one vaginal intercourse within the last three months
* Willing and able to give written informed consent (or if desired, consent provided by parent or guardian with written assent from the minor participant)
* Provide locator information to study staff throughout the trial
* Comply with all aspects of the study protocol, including random assignment to the Carraguard® plus condom or placebo plus condom arm, clinical valuations, specimen collection and testing, visit schedule and study drug regimen
* Citizen or permanent resident of South Africa
* Resident for the past year and intends to reside in the catchment area of the site for the next two years
* During the study, will not use any vaginal products except tampons or those prescribed or approved by the study clinician.

Exclusion Criteria:

* Currently pregnant, or indicate a desire to become pregnant in the next two years at the time of screening
* Within four weeks of last pregnancy outcome at the time of enrolment
* Pap smear at screening is graded as carcinoma.
* Injected illicit drugs in the 12 months prior to screening
* Participating in any other clinical trial/HIV prevention study

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6203 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Time to HIV seroconversion during trial participation (evaluated quarterly)

SECONDARY OUTCOMES:
Determine long-term safety based on the incidence of sexually transmitted infections (STI), Chlamydia, gonorrhoeae, trichomoniasis, and syphilis tests and the number of adverse events and serious adverse events
Chlamydia, gonorrhoeae, trichomoniasis and syphilis tests are conducted at months 3, 6, 12, 18 and 24 and as clinically indicated

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Lahteenmaki, MD, PhD, Principal Investigator — Population Council, Center for Biomedical Research
Locations (3):
- South Africa (3):
  - Isipingo Clinic, Overport, Durban
  - Empilisweni Clinic, Cape Town
  - Setshaba Research Clinic, University of Limpopo - Medunsa Campus, Medunsa

REFERENCES:
- [Background] Skoler S, Govender S, Altini L, Ahmed K, Waldron D, Myer L, Lahteenmaki P. Risks in the use of an unblinded-control group. J Infect Dis. 2005 Apr 15;191(8):1378-9; author reply 1379-80. doi: 10.1086/427833. No abstract available. PMID 15776387
- [Background] Wallace AR, Teitelbaum A, Wan L, Mulima MG, Guichard L, Skoler S, Vilakazi H, Mapula FS, Rossier J, Govender SN, Lahteenmaki P, Maguire RA, Phillips DM. Determining the feasibility of utilizing the microbicide applicator compliance assay for use in clinical trials. Contraception. 2007 Jul;76(1):53-6. doi: 10.1016/j.contraception.2006.10.012. Epub 2007 May 11. PMID 17586138
- [Background] Singh JA, Karim SS, Karim QA, Mlisana K, Williamson C, Gray C, Govender M, Gray A. Enrolling adolescents in research on HIV and other sensitive issues: lessons from South Africa. PLoS Med. 2006 Jul;3(7):e180. doi: 10.1371/journal.pmed.0030180. Epub 2006 Apr 18. PMID 16608384
- [Derived] Skoler-Karpoff S, Ramjee G, Ahmed K, Altini L, Plagianos MG, Friedland B, Govender S, De Kock A, Cassim N, Palanee T, Dozier G, Maguire R, Lahteenmaki P. Efficacy of Carraguard for prevention of HIV infection in women in South Africa: a randomised, double-blind, placebo-controlled trial. Lancet. 2008 Dec 6;372(9654):1977-87. doi: 10.1016/S0140-6736(08)61842-5. PMID 19059048
- See also: Official website of the Population Council — http://www.popcouncil.org